CLINICAL TRIAL: NCT01865734
Title: Comparison of Usual Podiatric Care and Early Physical Therapy for Plantar Heel Pain: A Randomized Clinical Trial
Brief Title: Comparison of Usual Podiatric Care and Early Physical Therapy for Plantar Heel Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Des Moines University (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 04-13-02
Record Dates: First submitted 2013-05-24; First posted 2013-05-31 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Fasciitis, Plantar
Keywords: Fasciitis, Plantar; Heel Pain; Physical Therapy; Podiatry; Musculoskeletal Manipulations; Exercise Therapy
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Physical Therapy (Experimental): Physical therapy after initial podiatry visit
  Interventions: Other: Physical therapy after initial podiatry visit
- Usual Podiatric Care (Active Comparator): Usual care provided by podiatry
  Interventions: Other: Usual care provided by podiatry

INTERVENTIONS:
Other: Physical therapy after initial podiatry visit — Individuals in the early physical therapy group will receive physical therapy in accordance with the American Physical Therapy Association plantar heel pain practice guidelines and recent evidence in support of manual therapy intervention. Treatment provided will be based on identified impairments and may include manual therapy (joint and soft tissue mobilization/thrust manipulation to the lower half of the body), lower leg and plantar foot specific stretching/self mobilization, foot and lower leg muscle performance training, night splints, taping, over the counter orthotics/heel cup/heel cushion, and iontophoresis. Specific intervention will be selected at the discretion of the treating physical therapist.
  Arms: Early Physical Therapy
Other: Usual care provided by podiatry — Individuals in the usual podiatric care group will receive care typical of podiatry management of plantar heel pain. According to practice guidelines, the first 6 weeks of treatment includes foot taping/padding, home stretching exercises, arch support/heel cup, shoe recommendations, oral anti-inflammatories, and corticosteroid injection. The next 6 months may include corticosteroid injection, custom orthotics, night splint, immobilization, and physical therapy. If unresponsive after 6 months of treatment, extracorporal shock wave therapy or a fasciotomy surgery is considered. Additionally, the podiatrist may order radiographs or ultrasound imaging within their scope of practice. Specific intervention will be selected at the discretion of the treating podiatrist.
  Arms: Usual Podiatric Care

SUMMARY:
Plantar heel pain (PHP) is one of the most common foot conditions in podiatry and physical therapy practice and often is associated with chronic symptoms, and disability. Persistence of symptoms adds to the economic burden of PHP and cost-effective solutions are needed to reduce this burden. Currently, there is wide variation in treatment, cost, and outcomes of care for PHP. Two practice guidelines are available to direct management patterns, but the guidelines and recent evidence of PHP interventions are unclear about the timing and influence of physical therapy in the multidisciplinary management of PHP. The purpose of this investigation is to compare the outcomes and costs associated with early physical therapy (ePT) following initial presentation to podiatry versus usual podiatric care (uPOD) in individuals with PHP. It is hypothesized that there will be greater improvement and/or reduced costs associated with either ePT or uPOD. In this study, 112 individuals with PHP will be randomized to receive uPOD or ePT after an initial visit with a podiatrist. Treatment provided in the uPOD group will reflect usual management patterns and intervention will be determined by the podiatrist. Treatment provided in the ePT group will be determined by the physical therapist and will focus on impairment-based manual therapy and exercise to the lower half of the body. In addition, evidence-based pain modulating modalities will be integrated into ePT treatment. Comparisons will be made between groups in the Foot and Ankle Ability measure (FAAM), the European Quality of Life (EQ-5D), Numeric Pain Rating Scale (NPRS), Global Rating of Change (GROC), and cost of treatment at 6, 26, and 52, weeks. The association between successful outcome based on GROC score and patient expectation of physical therapy or podiatry, and general expectations of symptom improvement will be analyzed. The results of this investigation will help to determine the impact of ePT to inform practice, update existing guidelines to reduce practice variation, and identify the most cost effective treatment for patients with PHP.

DETAILED DESCRIPTION:
This investigation will be a randomized clinical trial comparing participant-reported outcomes and cost-effectiveness of ePT and uPOD with follow up extending to 1 year. Following eligibility screening and completion of study questionnaires participants will be randomized using concealed envelopes and proceed with the intervention of their assigned group. Outcomes will be collected at 6 weeks, 6 months, and 1 year after initial presentation. All outcomes will be completed by the patient without any influence from investigators aware of the group assignment. Data entry and processing will occur by an investigator blinded to group allocation. A small financial incentive will be provided to facilitate completion of outcome measures over the study duration.

Statistical Analysis: Baseline group variables will be summarized using the mean and standard deviation for continuous measures and percentages for categorical measures. Independent t-tests (p<0.05, two-tailed) or the appropriate nonparametric test will be used to compare between group differences in baseline characteristics. Parametric test assumptions will be analyzed for all continuous variables by visual inspection of histograms, use of skewness score within double the standard error of skewness criteria, and Levene's test for homogeneity of the variance. A repeated measures analysis of variance will be used to compare group differences in the FAAM, NPRS, EQ-5D, and number of office visits associated with treatment at each time point. Results will be reported as the group mean, mean difference between groups, 95% confidence intervals, f-value, p-value, power, and effect size. The chi-square test will be used to compare GROC scores between groups at each time point and results will be reported as the chi-square value, p-value, and the frequency per category. The types of treatment based on Current Procedural Terminology (CPT) and Healthcare Common Procedure Coding System (HCPS) codes provided per group will be reported as percentages. Analysis of covariance will be used if any group differences are observed in participant characteristics. Intention to treat analysis will be performed by comparing the complete case analysis to multiple imputation analysis. Multiple imputed data sets will be generated using the Multivariate Imputation by Chained Equations algorithm with SPSS 19.0 for Windows (SPSS Inc., Chicago, IL, USA). Multinomial logistic regression will be used to obtain pooled regression estimates from the data sets which will be used for analysis. Post-randomization exclusion of included participants that did not meet eligibility criteria or that did not receive intervention will be considered for exclusion of the analysis by an independent, blinded adjudication committee that will evaluate all randomized participants. Any cross-overs will be analyzed in the original group they were assigned to and compared to an analysis that excludes cross-overs.

Participant expectations and preferences for ePT or uPOD will be categorized into 3 categories; matched, unmatched and neutral. Participants will be labelled 'matched' if they are allocated to a group for which they have expressed a higher expectation of benefit. A higher expectation will be denoted by comparison of visual analog ratings between the groups (ePT and uPOD). Unmatched participants will be those who are allocated to the treatment group for which they have a lower expectation of benefit. Neutral participants will be those who indicate the same level of expectation for both treatments. Similar categorizations will be made for participant preference based upon their response to the treatment preference question. General expectations of improvement will be dichotomized into met or unmet based upon rankings at the 6 week, 6 month, and 1 year follow-up relative to baseline rankings. Participants that demonstrate 6 week, 6 month, and 1 year ranks equal to or higher than baseline will be considered to have met their global expectations of improvement. Participants that demonstrate rankings below baseline expectations will be considered to have unmet global expectations of improvement. A chi-square test of independence will be used to compare the proportions of individuals with matched/unmatched/neutral expectations or preferences to global expectations (met or unmet). In addition, differences in expectation and preference categories will be analyzed relative to treatment success using a chi-square test of independence. Treatment success will be determined by the GROC at each time period with success defined as a GROC of +5, "a great deal better," or greater.

Power Analysis: Sample size estimates were calculated based on the primary outcome measure, the FAAM, at 6 months. In the absence of research comparing physical therapy and podiatry interventions or podiatry interventions using the FAAM as an outcome measure, sample size calculations were based on achieving a clinically meaningful difference between the groups and details from a recent clinical trial by Cleland et al that used similar methods to this investigation. Sample size estimate was made using G*Power 3.1.5 based on detecting a difference between groups greater than the minimal clinically important difference (MCID; ie, 9 point change) of the FAAM at 6 months with an alpha level of 0.05, 80% power, and pooled sample variance of 14.5 from Cleland et al This resulted in an effect size of 0.62 and 42 participants needed per group. This estimate is similar to the effect size of 0.69 achieved in the Cleland et al study that had 27 subjects per 2 treatment groups. To account for participants who drop-in or drop-out of treatment, in addition to the possibility of some participants not returning the FAAM questionnaire, the sample will be increased by 33% resulting in 56 participants per group. This estimate is conservative relative to the 3% drop-out rate and 7% rate of individuals that did not return outcome forms at the 6 month follow-up in the Cleland et al investigation. Significant effort will be made to retain subjects to include financial incentives and follow-up by the research assistant to assure completion and return of all outcome forms. The focus, and consequently the power analysis, of this investigation is on functional outcome (based on FAAM scores) and therefore may result in underpowered analysis of secondary variables.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Plantar Heel Pain: Tenderness to palpation of the plantar heel, pain associated with first step after waking, or pain with progression of daily weightbearing
* Patient's primary complaint is plantar heel pain

Exclusion Criteria:

* Score less than 74/84 on the Foot and Ankle Ability Measure activities of daily living (ADL) subscale
* Unable to complete questionnaires
* No treatment for heel pain in last 6 weeks
* Duration of symptoms greater than 1 year
* Current fracture of the lower leg, ankle, or foot
* Neurological condition affecting function of lower leg
* Advanced peripheral artery disease
* Rheumatoid arthritis
* Osteoporosis
* Active cancer
* Prolonged steroid use
* Surgery of the lower leg, ankle, or foot

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure | 6 months

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Baseline, 6 weeks, 6 months, 1 year
  The average of the least, current, and worst pain in the last week will be used.
Global Rating of Change Scale | 6 weeks, 6 months, 1 year
Incremental cost-effectiveness ratio | 6 weeks, 6 months, 1 year
  Incremental cost-effectiveness ratio will be calculated per quality-adjusted life year (QALY) gained determined by response on the European Quality of Life - 5 Dimensions
Foot and Ankle Ability Measure | Baseline, 6 weeks, and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shane McClinton, PT, DPT, Principal Investigator — Des Moines University
Locations (1):
- Des Moines University, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McClinton SM, Heiderscheit BC, McPoil TG, Flynn TW. Effectiveness of physical therapy treatment in addition to usual podiatry management of plantar heel pain: a randomized clinical trial. BMC Musculoskelet Disord. 2019 Dec 28;20(1):630. doi: 10.1186/s12891-019-3009-y. PMID 31883516
- [Derived] McClinton SM, Flynn TW, Heiderscheit BC, McPoil TG, Pinto D, Duffy PA, Bennett JD. Comparison of usual podiatric care and early physical therapy intervention for plantar heel pain: study protocol for a parallel-group randomized clinical trial. Trials. 2013 Dec 3;14:414. doi: 10.1186/1745-6215-14-414. PMID 24299257